CLINICAL TRIAL: NCT06485713
Title: Efficacy and Safety of Trifluridine/Tipiracil Combined With Fufuquitinib Versus Trifluridine/Tipiracil and Fufuquitinib for Third-line Treatment of Unresectable Metastatic Colorectal Cancer
Brief Title: Efficacy and Safety of Trifluridine/Tipiracil Combined With Fufuquitinib for Third-line Treatment of mCRC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KY2023-046
Record Dates: First submitted 2024-04-11; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Metastatic Colorectal Cancer; Drug Therapy
Keywords: Metastatic Colorectal Cancer; Fufuquitinib; trifluridine/tipiracil; Combination therapy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Trifluridine; trifluridine tipiracil drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Experimental group (Experimental): trifluridine/tipiracil combined with fufuquitinib
  Interventions: Drug: trifluridine/tipiracil combined with fufuquitinib
- Control Group 1 (Active Comparator): Fufuquitinib
  Interventions: Drug: fufuquitinib
- Control Group 2 (Active Comparator): Trifluridine/tipiracil
  Interventions: Drug: Trifluridine/tipiracil

INTERVENTIONS:
Drug: trifluridine/tipiracil combined with fufuquitinib — trifluridine/tipiracil combined with fufuquitinib
  Arms: Experimental group
Drug: fufuquitinib — fufuquitinib
  Arms: Control Group 1
Drug: Trifluridine/tipiracil — Trifluridine/tipiracil
  Arms: Control Group 2

SUMMARY:
To evaluate the efficacy and safety of trifluridine/tipiracil combined with fufuquitinib versus trifluridine/tipiracil and fufuquitinib in patients with unresectable metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1.Age 18-75 (at the time of signing the informed consent);ECOG PS score: 0-1; Expected survival time > 3 months.

  2.Patients with advanced colorectal adenocarcinoma confirmed by histopathology who had failed standard first - and second-line treatment.

  3.At least 1 measurable lesion was present according to RECIST1.1 criteria. 4.Good organ function, laboratory tests meet the following criteria:
  1. Hemoglobin ≥90g/L;Absolute count of neutrophils (ANC) ≥1.5×109/L;Platelet ≥100×109/L;
  2. ALT and AST≤2.5 upper limit of normal (ULN).ALP≤2.5 ULN;(if liver metastases ≤5 ULN);
  3. Total bilirubin (TBIL) < 1.5 ULN;
  4. Serum creatinine (CR) <1.5 ULN or creatinine clearance (CCR) ≥50ml/min;
  5. Serum albumin ≥30g/L;
  6. International Normalized ratio (INR), prothrombin time (PT), activated partial thrombin time (APTT) ≤1.5ULN;
  7. Thyrotropin (TSH) ≤ULN;If abnormal, T3 and T4 levels should be investigated, and normal levels can be included.

     5.cardiac color ultrasound: Left ventricular ejection fraction (LVEF) ≥50%. 6.Hypertension was well controlled. 7.Female participants of reproductive age should agree to use contraception during the study period and for 6 months after the study ends; Serum pregnancy test was negative within 7 days prior to study enrollment,and should be Non-lactation stage. Male subjects should agree to use contraception during the study period and for 6 months after the study ends.

     Exclusion Criteria:
* 1.Combined disease or history

  1. .Present or present with other malignancies within 3 years.
  2. .Have multiple factors affecting oral medication (such as inability to swallow, chronic diarrhea, or intestinal obstruction)
  3. .Gastrointestinal bleeding or perforation occurred during the first 4 weeks of enrollment
  4. .Patients with ulcerative colitis, Crohn's disease, and active inflammatory bowel disease during the first 4 weeks of enrollment
  5. .Uncontrolled pleural effusion, ascites, and moderate or greater pericardial effusion
  6. .Unmitigated toxic reactions above grade 1 of CTC AE due to any previous treatment, excluding alopecia.
  7. .Received major surgical treatment or significant traumatic injury within 28 days prior to enrollment
  8. .Patients with hematemesis, hematochezia, or any bleeding event ≥ CTCS AE level 3 within the previous 3 months, or with any signs of bleeding or history determined by the investigator to be ineligible for enrollment
  9. .Arteriovenous thrombosis occurred within 6 months, such as cerebrovascular accident, pulmonary embolism, etc
  10. .A history of psychotropic substance abuse and inability to abstain
  11. .Subjects with any severe and/or uncontrolled disease, including

      1. Uncontrolled hypertension
      2. Unstable angina pectoris / ≥ grade 2 cardiogenic chest pain;Myocardial infarction occurred within 12 months before randomization;≥ grade 2 heart failure;Restrictive heart disease;≥ grade 2 atrioventricular block, arrhythmia that cannot be stably controlled with drugs.
      3. Active infection
      4. Decompensated cirrhosis, active hepatitis;
      5. Renal failure requires hemodialysis or peritoneal dialysis
      6. A history of immunodeficiency, including HIV positive or other acquired, congenital immunodeficiency diseases, or a history of organ transplantation

      h.Diabetes with poorly controlled i.Urine routine showed urine protein ≥++, and 24h albuminuria quantitative > 1.0 g g.History of neurological or psychiatric disorders 2.Subjects who, in the investigator's judgment, have a concomitant medical condition that seriously endangers subjects' safety or interferes with the completion of the study, or are deemed unsuitable for enrollment for other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | up to 24 weeks

SECONDARY OUTCOMES:
Total survival time | up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Quasar Collaborative Group; Gray R, Barnwell J, McConkey C, Hills RK, Williams NS, Kerr DJ. Adjuvant chemotherapy versus observation in patients with colorectal cancer: a randomised study. Lancet. 2007 Dec 15;370(9604):2020-9. doi: 10.1016/S0140-6736(07)61866-2. PMID 18083404
- [Background] Twelves C, Wong A, Nowacki MP, Abt M, Burris H 3rd, Carrato A, Cassidy J, Cervantes A, Fagerberg J, Georgoulias V, Husseini F, Jodrell D, Koralewski P, Kroning H, Maroun J, Marschner N, McKendrick J, Pawlicki M, Rosso R, Schuller J, Seitz JF, Stabuc B, Tujakowski J, Van Hazel G, Zaluski J, Scheithauer W. Capecitabine as adjuvant treatment for stage III colon cancer. N Engl J Med. 2005 Jun 30;352(26):2696-704. doi: 10.1056/NEJMoa043116. PMID 15987918
- [Background] Yothers G, O'Connell MJ, Allegra CJ, Kuebler JP, Colangelo LH, Petrelli NJ, Wolmark N. Oxaliplatin as adjuvant therapy for colon cancer: updated results of NSABP C-07 trial, including survival and subset analyses. J Clin Oncol. 2011 Oct 1;29(28):3768-74. doi: 10.1200/JCO.2011.36.4539. Epub 2011 Aug 22. PMID 21859995